CLINICAL TRIAL: NCT03116490
Title: The Comparative Effects of Regional or General Anesthesia on the Prognosis of Hip Fracture Surgery on Elderly Patients
Brief Title: The Effects of Anesthesia Type on the Prognosis of Hip Fracture Surgery on Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Ting Li, Director,Associate chief physician of Anesthesia Department, Wenzhou Medical University
Other Study IDs: RAGA-PHP
Record Dates: First submitted 2017-01-14; First posted 2017-04-17 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Complications; Postoperative Mortality
Keywords: morbidity; mortality; hip fracture; anesthesia type; POSSUM
MeSH Terms: conditions — Postoperative Complications; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group RA: the anesthesia type for patients with hip fracture surgery is regional anesthesia
  Interventions: Procedure: Anesthesia type
- group GA: the anesthesia type for patients with hip fracture surgery is general anesthesia
  Interventions: Procedure: Anesthesia type

INTERVENTIONS:
Procedure: Anesthesia type — RA group uses regional anesthesia(epidural, spinal, combined spinal and epidural anesthesia or nerve block) ,and GA group uses general anesthesia(general anesthesia combined with peripheral nerve blockade, general anesthesia combined with spinal/epidural anesthesia or single general anesthesia) .

SUMMARY:
The aim of this study is to figure out whether anesthesia type have an influence on the prognosis of hip fracture surgery.30-day mortality and morbidity after the surgery are our main observational index,and according to literature and our experience,regional anesthesia may have a better prognosis after hip fracture surgery compared with general anesthesia.

DETAILED DESCRIPTION:
Hip fracture is a common disease among elderly people,and has a high mortality and morbidity.But,seldom practice can be done to improve this condition.For a long time,whether anesthesia type could influence the prognosis after surgery is controversial.Several studies have confirmed regional anesthesia may be better for patients for its fewer complications.But most studies are retrospective,and information may be less convincing .Besides,as a matter of fact,patients of different anesthesia type may have different status,so,a scoring system may be need for comparing the status of patients of different groups.

Our study is a prospective observational trial.Patients needing hip fracture surgery are divided into two groups according to the anesthesia type during surgery:Regional Anesthesia group(RA),General Anesthesia group(GA).To evaluate the status of patients before surgery,we use Orthopedic POSSUM scoring system.It consists of 12 physiological factors and 6 operative severity factors.Then,we will observe outcome of the two groups and record every complication after surgery.Finally,the initial and adjusted morbidity and mortality according to Orthopedic POSSUM scoring system of the two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fracture;
* Need surgery;
* Anesthesia type is regional anesthesia or general anesthesia;
* Age≥60 years.

Exclusion Criteria:

* Choosing conservative treatment;
* Other types of anesthesia or without anesthesia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients experiencing hip fracture surgery.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day after surgery

SECONDARY OUTCOMES:
Morbidity | 30-day after surgery
VAS pain score | everyday after surgery,record for 7 days

OTHER OUTCOMES:
The Orthopedic POSSUM score | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, M.D., Study Chair — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University; Yahe Ge, Medical Student, Principal Investigator — The Second Affiliated Hospital & Yuying Children hospital of Wenzhou Medical University
Locations (1):
- WenZhou Medical University Second Affiliated Hospital, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Radcliff TA, Henderson WG, Stoner TJ, Khuri SF, Dohm M, Hutt E. Patient risk factors, operative care, and outcomes among older community-dwelling male veterans with hip fracture. J Bone Joint Surg Am. 2008 Jan;90(1):34-42. doi: 10.2106/JBJS.G.00065. PMID 18171955
- [Background] Johnell O, Kanis JA. An estimate of the worldwide prevalence and disability associated with osteoporotic fractures. Osteoporos Int. 2006 Dec;17(12):1726-33. doi: 10.1007/s00198-006-0172-4. Epub 2006 Sep 16. PMID 16983459
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Parker M, Johansen A. Hip fracture. BMJ. 2006 Jul 1;333(7557):27-30. doi: 10.1136/bmj.333.7557.27. No abstract available. PMID 16809710
- [Background] Beaupre LA, Jones CA, Saunders LD, Johnston DW, Buckingham J, Majumdar SR. Best practices for elderly hip fracture patients. A systematic overview of the evidence. J Gen Intern Med. 2005 Nov;20(11):1019-25. doi: 10.1111/j.1525-1497.2005.00219.x. PMID 16307627
- [Background] Neuman MD, Archan S, Karlawish JH, Schwartz JS, Fleisher LA. The relationship between short-term mortality and quality of care for hip fracture: a meta-analysis of clinical pathways for hip fracture. J Am Geriatr Soc. 2009 Nov;57(11):2046-54. doi: 10.1111/j.1532-5415.2009.02492.x. Epub 2009 Sep 28. PMID 19793159
- [Background] Vestergaard P, Rejnmark L, Mosekilde L. Loss of life years after a hip fracture. Acta Orthop. 2009 Oct;80(5):525-30. doi: 10.3109/17453670903316835. PMID 19916683
- [Background] Vochteloo AJ, Borger van der Burg BL, Roling MA, van Leeuwen DH, van den Berg P, Niggebrugge AH, de Vries MR, Tuinebreijer WE, Bloem RM, Nelissen RG, Pilot P. Contralateral hip fractures and other osteoporosis-related fractures in hip fracture patients: incidence and risk factors. An observational cohort study of 1,229 patients. Arch Orthop Trauma Surg. 2012 Aug;132(8):1191-7. doi: 10.1007/s00402-012-1520-9. Epub 2012 Apr 24. PMID 22526197
- [Background] Parker MJ, Handoll HH, Griffiths R. Anaesthesia for hip fracture surgery in adults. Cochrane Database Syst Rev. 2001;(4):CD000521. doi: 10.1002/14651858.CD000521. PMID 11687085
- [Background] O'Hara DA, Duff A, Berlin JA, Poses RM, Lawrence VA, Huber EC, Noveck H, Strom BL, Carson JL. The effect of anesthetic technique on postoperative outcomes in hip fracture repair. Anesthesiology. 2000 Apr;92(4):947-57. doi: 10.1097/00000542-200004000-00011. PMID 10754613
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Neuman MD, Rosenbaum PR, Ludwig JM, Zubizarreta JR, Silber JH. Anesthesia technique, mortality, and length of stay after hip fracture surgery. JAMA. 2014 Jun 25;311(24):2508-17. doi: 10.1001/jama.2014.6499. PMID 25058085
- [Background] Patorno E, Neuman MD, Schneeweiss S, Mogun H, Bateman BT. Comparative safety of anesthetic type for hip fracture surgery in adults: retrospective cohort study. BMJ. 2014 Jun 27;348:g4022. doi: 10.1136/bmj.g4022. PMID 24972901
- [Background] Owens WD, Felts JA, Spitznagel EL Jr. ASA physical status classifications: a study of consistency of ratings. Anesthesiology. 1978 Oct;49(4):239-43. doi: 10.1097/00000542-197810000-00003. PMID 697077
- [Background] Copeland GP, Jones D, Walters M. POSSUM: a scoring system for surgical audit. Br J Surg. 1991 Mar;78(3):355-60. doi: 10.1002/bjs.1800780327. PMID 2021856
- [Background] Brunelli A, Fianchini A, Xiume F, Gesuita R, Mattei A, Carle F. Evaluation of the POSSUM scoring system in lung surgery. Physiological and Operative Severity Score for the enUmeration of Mortality and Morbidity. Thorac Cardiovasc Surg. 1998 Jun;46(3):141-6. doi: 10.1055/s-2007-1010211. PMID 9714489
- [Background] Gotohda N, Iwagaki H, Itano S, Horiki S, Fujiwara T, Saito S, Hizuta A, Isozaki H, Takakura N, Terada N, Tanaka N. Can POSSUM, a scoring system for perioperative surgical risk, predict postoperative clinical course? Acta Med Okayama. 1998 Dec;52(6):325-9. doi: 10.18926/AMO/31304. PMID 9876770
- [Background] Tekkis PP, Kocher HM, Bentley AJ, Cullen PT, South LM, Trotter GA, Ellul JP. Operative mortality rates among surgeons: comparison of POSSUM and p-POSSUM scoring systems in gastrointestinal surgery. Dis Colon Rectum. 2000 Nov;43(11):1528-32, discusssion 1532-4. doi: 10.1007/BF02236732. PMID 11089587
- [Background] Mohamed K, Copeland GP, Boot DA, Casserley HC, Shackleford IM, Sherry PG, Stewart GJ. An assessment of the POSSUM system in orthopaedic surgery. J Bone Joint Surg Br. 2002 Jul;84(5):735-9. doi: 10.1302/0301-620x.84b5.12626. PMID 12188495
- [Background] Wright DM, Blanckley S, Stewart GJ, Copeland GP. The use of orthopaedic POSSUM as an audit tool for fractured neck of femur. Injury. 2008 Apr;39(4):430-5. doi: 10.1016/j.injury.2007.11.009. Epub 2008 Mar 7. PMID 18316084
- [Background] OVERALL JE, WILLIAMS CM. Models for medical diagnosis. Behav Sci. 1961 Apr;6:134-41. doi: 10.1002/bs.3830060205. No abstract available. PMID 13731759